CLINICAL TRIAL: NCT01770197
Title: The Feasibility and Outcome of Intravenous Thrombolysis for Stroke Patients in the 3-4.5 Hour Time Window in China
Brief Title: Outcome of Intravenous Thrombolysis for Stroke Patients in the 3-4.5 Hour Time Window
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, zhipeng xu, Wuhan General Hospital of Guangzhou Military Command, Wuhan General Hospital of Guangzhou Military Command
Other Study IDs: 20090101
Record Dates: First submitted 2013-01-08; First posted 2013-01-17 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Stroke
Keywords: China; Stroke; Thrombolytic therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- recombinant tissue plasminogen activator: Stroke patients with rt-PA treatment in the 3-4.5 hour time window were compared with those within 3h.
  Interventions: Drug: IV rt-PA
- rt-PA: One group of was treated with standard recombinant tissue plasminogen activator therapy in 3h and the other group of stroke patients was treated within 3-4.5h.
  Interventions: Drug: IV rt-PA

INTERVENTIONS:
Drug: IV rt-PA — IV rt-PA treatment
  Other Names: rt-PA

SUMMARY:
The time window for intravenous recombinant tissue plasminogen activator treatment in ischemic stroke patients has been extended to 4.5h. Little is known about intravenous recombinant tissue plasminogen activator use in the 3-4.5 hour time window among Chinese stroke patients. This exploratory study was to describe the feasibility and outcome of treatment with intravenous recombinant tissue plasminogen activator in the expanded time window, and to offer suggestions for future clinical work in China.

DETAILED DESCRIPTION:
Favorable clinical outcome of intravenous recombinant tissue plasminogen activator was assessed by absolute changes in the National Institute of Health Stroke Scale score at 24 hours and by the improvement of modified Rankin Scale score at discharge or 6-month follow-up. The safety of intravenous recombinant tissue plasminogen activator was assessed by the rate of mortality, intracerebral hemorrhage and other common complications. Multivariate logistic regression models were used to evaluate factors associated with favorable clinical outcome.

ELIGIBILITY:
Inclusion Criteria:stroke patients in the 3-4.5 hour time window -

Exclusion Criteria:stroke patients in more than 4.5 hour time window

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients in the 3-4.5 hour time window
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
National Institute of Health Stroke Scale score and modified Rankin Scale | Outcome measure will be assessed at 24 weeks
  Favorable clinical outcome of intravenous recombinant tissue plasminogen activator was assessed by absolute changes in the National Institute of Health Stroke Scale score at 24 hours and by the improvement of modified Rankin Scale score at discharge or 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wuhan G H, High, Study Chair — Wuhan General Hospital of Guangzhou Command

REFERENCES:
- See also: Outcome of Intravenous Thrombolysis for Stroke Patients in the 3-4.5 Hour Time Window — http://ClinicalTrials.gov